CLINICAL TRIAL: NCT03488498
Title: Multicenter Investigation Weight Bath Traction in Chronic Lumbar Spine Pain: a Controlled, Randomiezd, Single Blind Follow-up Study
Brief Title: Weight Bath Traction in Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: Polyclinic of the Hospitaller Brothers of St. John of God, Budapest (Other)
Responsible Party: Principal Investigator, Tamas Gati, Principal Investigator, Polyclinic of the Hospitaller Brothers of St. John of God, Budapest
Other Study IDs: 21396-3/2017/EKU
Record Dates: First submitted 2018-02-26; First posted 2018-04-05 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Low Back Pain
Keywords: Balneotherapy; Chronic low back pain; Controlled; Randomized trial; weight bath traction; follow-up
MeSH Terms: conditions — Low Back Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Receiving NSAID medication: Receiving NSAID medication
  Interventions: Other: questionnaires
- Receiving NSAID medication and weight bath therapy,
  Interventions: Other: questionnaires
- Receiving weight bath therapy,
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — Examination of the spinal mobilization in cm. The pain and quality of life assessment of functional status through questionnaires.

SUMMARY:
It is typical of chronic low back pain that, after the first painful episode, is repeated at 44-78% of patients. For acute lumbar pain, approx. 10-15% of them are converted into chronic. Conservative treatments are few studies done in the traction therapy. A large number of multicenter trials did not evaluate the effectiveness of underwater traction therapy.

DETAILED DESCRIPTION:
Goals are the followings:

1. Is the beneficial effect of a weight bath comparable to a non-treated control group with respect to clinical parameters?
2. How much does the quality of life change in an initial state and how much is it in comparison with the control group?

ELIGIBILITY:
Inclusion Criteria:

* at least 12 weeks of non-specific lymphatic pain,
* the pain sensitivity of the paravertebral muscle and the painful movement of the lumbar spine can be observed, which can be characterized by segmental motion, segmental instability or other reasons
* radiographically confirmed spondylosis, discopathy, and spondylarthrosis within one year.
* back pain at least 30mm (100mm visualis analogue scale).
* patients could not received systemic or locally administered steroid therapy, physiotherapy or they get balneotherapy in the last 2 months

  p- atient consent form signed before the start of test

Exclusion Criteria:

* The exclusion criteria included previous lumbar spine surgery,
* progressive neurologic loss,
* pregnancy,
* (umbilical, hiatal, inguinal) hernia,
* malignities,
* infectious diseases,
* inflammatory pathologies,
* severe pulmonary and cardiovascular diseases,
* uncontrolled- hypertension,
* mental disorders,
* incontinence,
* Acute lower back pain;
* Organic neurological symptoms associated with the lower back;
* pain in the background of osteoporosis or other causes of vertebral compression is likely
* Lack of complience,
* Pain due to inflammatory spinal disease;
* spondylolisthesis (which is not greater than 25% of vertebral skeleton compared to adjacent vertebrae)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are selected from on the Outpatients clinics of the Department of Rheumatology and Physiotherapy of Polyclinic of the Hospitaller Brothers of St. John of God, Budapest
Sampling Method: Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
prove the hypothesis that weight bath traction has favorable effect. of LBP using the change in the clinical parameters. | at the first visit and After at the 3 and the 12 weeks
  Change From Baseline in Pain Scores on the Visual Analog Scale at the 3 and the 12 weeks after the treatment.Pain intensity was measured by using the Visual Analog Scale (0-100 mm). Patients recorded on the VAS scale the level of low back pain at rest as well as during activity.

SECONDARY OUTCOMES:
Secondary objective was to evaluate whether it also leads to the improvement in the quality of life. | at the first visit and After at the 3 and the 12 weeks
  Change From Baseline in level of disability in 10 everyday activities of daily life , the Functional disability by using the Oswestry Disability Index (ODI) .
Secondary objective was to evaluate whether it also leads to the improvement in the quality of life. | at the first visit and After at the 3 and the 12 weeks
  the EuroQol Five Dimensions Questionnaire (EQ-5D). A self administered questionnaire instrument for measuring generic health status (health-related quality of life).
Secondary objective was to evaluate whether it also leads to the improvement in the movements of the lumbal spine. | at the first visit and After at the 3 and the 12 weeks
  Change From Baseline in level improvements in the parameters of clinical lumbal spine movements in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Tamas GATI, MD, Principal Investigator — Polyclinic of the Hospitaller Brothers of St. John of God,
Locations (1):
- Polyclinic of the Hospitaller Brothers of St. John of God,, Budapest, Árpád Fejedelem Útja 7, Hungary

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gati T, Czimer E, Cserhati G, Feher J, Olah M, Kulisch A, Mando Z, Bender T. A multicentre randomized controlled follow-up study of the effects of the underwater traction therapy in chronic low back pain. Int J Biometeorol. 2020 Aug;64(8):1393-1400. doi: 10.1007/s00484-020-01919-8. Epub 2020 May 2. PMID 32361959